CLINICAL TRIAL: NCT00874133
Title: The Effect of Acupuncture on Symptoms, Gastric Emptying Rate and Glucose Control in Patients With Diabetic Gastroparesis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Completed due to low number of eligible patients
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, dickman ram, MD, Rabin Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 004589
Record Dates: First submitted 2009-03-25; First posted 2009-04-02 (Estimated); Last update posted 2013-12-06 (Estimated); Status verified 2013-12

CONDITIONS: Diabetic Gastroparesis
MeSH Terms: interventions — Acupuncture Therapy; Domperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Motillium (Active Comparator): 20 mg motilium thrice daily for 12 weeks.
  Interventions: Drug: Motilium
- Acupuncture (Active Comparator): Acupuncture treatment.
  Interventions: Procedure: Acupuncture

INTERVENTIONS:
Procedure: Acupuncture — Acupuncture treatment for 12 weeks.
  Other Names: Domperidone
  Arms: Acupuncture
Drug: Motilium — 20 mg motilium thrice daily
  Other Names: Domperidone
  Arms: Motillium

SUMMARY:
Diabetes affects 5.8% of the adult population in Israel (1). Gastroparesis is a syndrome characterized by delayed gastric emptying in the absence of mechanical obstruction of the stomach.Treatment with acupuncture has been described as effective in improvement of symptoms in patients with gastroparesis in a number of patient series. However, this treatment approach has not been tested by means of a controlled randomized clinical study, and neither has the connection between improvement of symptoms and the anatomical-physiological effect of the treatment, if ever, assessed.This study will test the efficacy of motilium (20 mg thrice daily) as compared to acupuncture treatment on the following subjective and objective parameters of 30 patients with diabetic gastroparesis and impaired glucose control:

1. To compare the degree of GCSI scores improvement before and after treatment with motilium or acupuncture using a validated questionnaire.
2. To determine the effect of treatment with motilium or acupuncture on gastric emptying rate.
3. To determine the effect of treatment with motilium or acupuncture on glycemic control.
4. To compare the quality of life before and after treatment with motilium or acupuncture using the Short Form-36 (SF-36).

DETAILED DESCRIPTION:
This is a randomized, comparative, pilot study, which will compare two treatments: acupuncture treatment vs. treatment with motilium in 30 diabetic patients with impaired glucose control and gastroparesis.

All patients who meet inclusion criteria will undergo gastric scintigraphy and upper endoscopy to assess the presence of gastroparesis and to rule out gastric outlet obstruction. At baseline, all enrolled patients will fill out the Gastroparesis Cardinal Symptom Index (GCSI), the Quality of life questionnaire (SF-36). Subsequently, patients will be randomized to 20 mg motilium thrice daily and after 1 month wash-out period to acupuncture treatment, each treatment will last 12 weeks.

After treatment, patients will undergo a second gastric scintigraphy and will complete the GCSI and the SF-36.

Fasting blood glucose concentrations and HbA1c levels will be determined at the beginning and at the end of the study and at 6 months later as well.

End Points:

Primary: Level of improvement of gastric emptying rate, and improvement in blood glucose levels at the end of treatment, in comparison with tests before treatment.

Secondary: Level of improvement in scores of severity of gastroparesis related symptoms, with quality of life indicators, in comparison with tests before treatment; also, the number of visits to family doctors/diabetic clinics/emergency rooms, as well as use of the medications resulting from diabetic complications will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-80,
* Diabetic patients of over 10 years duration with impaired glucose control, after at least 6 months of accepted treatment in a Diabetes Clinic by the study staff before inclusion in the study, who exhibit symptoms which could signify the possibility of diabetic gastroparesis.

Exclusion Criteria:

* Known hyperprolactinemia, systemic or localized neurological disturbances (myopathy, multiple sclerosis, Parkinson's disease, myelopathy), with the exception of diabetic neuropathy, past stomach or esophagus surgery, pregnancy, inability to sign Informed Consent, fear of acupuncture, limb amputation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2009-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Level of improvement of gastric emptying rate | 6 months

SECONDARY OUTCOMES:
Improvement in blood glucose levels | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ram Dickman, MD, Principal Investigator — RMC